CLINICAL TRIAL: NCT05748379
Title: Closure of a Guided Immediate Implant Placed in the Extraction Socket With Bone Augmentation in the Lateral Area of the Maxilla or Mandible, With a Temporary Composite Abutment vs With a Custom-made Zirconium Oxide Abutment.
Brief Title: Atraumatic Zirconia Abutment Versus Customized Composite Healing Abutment in Maxilla or Mandible.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SIA Adenta (Other)
Responsible Party: Principal Investigator, Vitālijs Gnusins, Doctor of dental Surgery, SIA Adenta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SIAAdenta
Record Dates: First submitted 2023-01-11; First posted 2023-02-28 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Dental Implants; Humans; Dental Implants, Single-Tooth; Male; Female; Osseointegration; Dental Anxiety; Guided Surgery

STUDY DESIGN:
Who Masked: Participant
Masking Description: Each patient has their individual ID number
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kompozite closure (Other): Immediate implant placement and temporary closure of tapered implants with a custom-made composite shaper after tooth extraction with bone augmentation by using allogeneic bone.
  Interventions: Procedure: Kompozite closure
- Individual abutment (Other): Immediate implant placement and temporary closure of tapered implant with a custom-made zirconium oxide abutment after tooth extraction with bone augmentation by using allogeneic bone.
  Interventions: Procedure: Individual abutment

INTERVENTIONS:
Procedure: Kompozite closure — Immediate implant placement and temporary closure of tapered implants with a custom-made composite shaper.
  Arms: Kompozite closure
Procedure: Individual abutment — Immediate implant placement and temporary closure of tapered implant with a custom-made zirconium oxide abutment.
  Arms: Individual abutment

SUMMARY:
40 patients are included in the study, 20 patients in group 1 (=closure with composite material shaper; test group) and 20 patients in group 2 (=closure with custom-made zirconia oxide abutment; control group).

Randomisation envelopes will be used for randomisation. Device under study: Straumann BLX, Roxolid® , SLActive® dental implants with a diameter of 3.5, 3.75, 4, 4.5 mm are used.

Allogenic bone botiss maxgraft® cortical granules are used as graft material.

Inclusion criteria:

1. Males and females at least 18 years of age or older.
2. One implant per patient.
3. Prior to any study-related activity, the subject must voluntarily sign informed consent, be willing and able to attend scheduled follow-up visits, and agree to the collection and analysis of pseudonymised data.
4. Lateral individual teeth (premolars and molars).
5. Class I extraction socket (intact buccal wall) or class II (1/3 of buccal wall).
6. The gingival contour of the tooth to be extracted - without recession.
7. Adjacent anterior teeth have no periodontal loss.
8. There are no implants in the adjacent teeth.
9. Non-traumatic tooth extraction, which results in intact walls of the socket.

Exclusion criteria:

1. Deep occlusion (severe, class II).
2. The patient smokes a lot (more than 10 cigarettes per day).
3. Systemic disease (osteoporosis).
4. No initial stability has been achieved after the implant insertion procedure.

DETAILED DESCRIPTION:
General Notes

40 patients are included in the study, 20 patients in group 1 (=closure with composite material shaper; test group) and 20 patients in group 2 (=closure with custom-made zirconia oxide abutment; control group).

Randomisation envelopes will be used for randomisation. Device under study: Straumann BLX, Roxolid® , SLActive® dental implants with a diameter of 3.5, 3.75, 4, 4.5 mm are used.

Allogenic bone botiss maxgraft® cortical granules are used as graft material.

Inclusion criteria:

1. Males and females at least 18 years of age or older.
2. One implant per patient.
3. Prior to any study-related activity, the subject must voluntarily sign informed consent, be willing and able to attend scheduled follow-up visits, and agree to the collection and analysis of pseudonymised data.
4. Lateral individual teeth (premolars and molars).
5. Class I extraction socket (intact buccal wall) or class II (1/3 of buccal wall).
6. The gingival contour of the tooth to be extracted - without recession.
7. Adjacent anterior teeth have no periodontal loss.
8. There are no implants in the adjacent teeth.
9. Non-traumatic tooth extraction, which results in intact walls of the socket.

Exclusion criteria:

1. Deep occlusion (severe, class II).
2. The patient smokes a lot (more than 10 cigarettes per day).
3. Systemic disease (osteoporosis).
4. No initial stability has been achieved after the implant insertion procedure. 4.2. Surgical Procedures and Recovery Phase (see Annexes No. 1 and 2)

Group 1. Immediate implant placement and temporary closure of tapered implants with a custom-made composite shaper after tooth extraction with bone augmentation by using allogeneic bone.

1. Non-traumatic extraction.
2. Palatal position of tapered implant for premolars and centred position for molars (more commonly - in the septum) 3-4 mm below the buccal gum line or 1-2 mm below the bony protuberance.
3. For premolars, the implant is placed palatally 2-3 mm to the buccal bone wall, for molars 2-3 mm to the buccal and lingual wall.
4. Implant insertion.
5. "Jump distance" sealing with allogeneic bone.
6. Temporary closure with a composite shaper.
7. Cone beam computed tomography with Carestream machine.
8. Taking a photo.
9. Scan with 3Shape TRIOS4 scanner.

After 3 months, a cone beam computed tomography is performed to evaluate changes in the crestal bone, the temporary restoration is screwed off and the presence/absence of bleeding is recorded. A digital impression is taken for a zirconium oxide crown made on Ti base and to assess soft tissue changes.

The change in the buccal vertical bone level will be measured as the difference between the former and the new vertical distance from implant platform to the buccal alveolar crest.

While the change in the buccal horizontal bone dimension will be measured as the difference between the former and the new horizontal distance between the implant and the outer surface of the buccal plate. Both measurements will be taken using CBCT, one immediately after the surgery and the other one 3 month later.

Intraoral scans with 3Shape Trios4 dental scanner will be taken to compare soft tissue stability. Measurements will be taken before, immediately after the surgery and 3 month later. By using STL files it will be possible to compare soft tissue stability.

Group 2. Immediate implant placement and temporary closure of tapered implant with a custom-made zirconium oxide abutment after tooth extraction with bone augmentation by using allogeneic bone.

1. Non-traumatic extraction.
2. Palatal position of tapered implant for premolars and centred position for molars (more commonly - in the septum) 3-4 mm below the buccal gum line or 1-2 mm below the bony protuberance.
3. For premolars, the implant is placed palatally 2-3 mm to the buccal bone wall, for molars 2-3 mm to the buccal and lingual wall.
4. Implant insertion.
5. "Jump distance" sealing with allogeneic bone.
6. Closure with a zirconium oxide abutment.
7. Cone beam computed tomography with Carestream machine.
8. Taking a photo.
9. Scan with 3Shape TRIOS4 scanner.

After 3 months, a cone beam computed tomography is performed to evaluate changes in the crestal bone, the custom-made abutment is screwed off and the presence/absence of bleeding is recorded. A digital impression is taken for a zirconium oxide crown and to assess soft tissue changes.

The change in the buccal vertical bone level will be measured as the difference between the former and the new vertical distance from implant platform to the buccal alveolar crest.

While the change in the buccal horizontal bone dimension will be measured as the difference between the former and the new horizontal distance between the implant and the outer surface of the buccal plate. Both measurements will be taken using CBCT, one immediately after the surgery and the other one 3 month later.

Intraoral scans with 3Shape Trios4 dental scanner will be taken to compare soft tissue stability. Measurements will be taken before, immediately after the surgery and 3 month later. By using STL files it will be possible to compare soft tissue stability.

Evaluation Phase

T1 (Basic): After the performance of final restoration: X-ray, photograph, scan, PD, BOP, RI.

T2: Follow-up after 3 months: X-ray, photograph, scan, PD, BOP, RI. T3: Follow-up after a year: X-ray, photograph, scan, PD, BOP, RI.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 18 years of age or older.
2. One implant per patient.
3. Prior to any study-related activity, the subject must voluntarily sign informed consent, be willing and able to attend scheduled follow-up visits, and agree to the collection and analysis of pseudonymised data.
4. Lateral individual teeth (premolars and molars).
5. Class I extraction socket (intact buccal wall) or class II (1/3 of buccal wall).
6. The gingival contour of the tooth to be extracted - without recession.
7. Adjacent anterior teeth have no periodontal loss.
8. There are no implants in the adjacent teeth.
9. Non-traumatic tooth extraction, which results in intact walls of the socket.

Exclusion Criteria:

1. Deep occlusion (severe, class II).
2. The patient smokes a lot (more than 10 cigarettes per day).
3. Systemic disease (osteoporosis).
4. No initial stability has been achieved after the implant insertion procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2025-05-22 (Estimated)

PRIMARY OUTCOMES:
Stability of crestal bone | Before surgery, immediately after surgery, 3 moth, 1 year follow up
  To compare crystal bone stability CBCT will be taken before surgery. , immediately after surgery, after 3 month and a follow up after 1 year.
  The change in the buccal vertical bone level will be measured as the difference between the former and the new vertical distance from implant platform to the buccal alveolar crest.
  While the change in the buccal horizontal bone dimension will be measured as the difference between the former and the new horizontal distance between the implant and the outer surface of the buccal plate. Both measurements will be taken using CBCT, one immediately after the surgery and the other one 3 month later
The changes of stability of soft tissue | Before surgery, immediately after surgery, 3 month, 1 year follow up
  Recession (REC) state of the gingival/mucosa border - registered by means of a periodontal probe from the incisal edge to the border of the medial, zenith and distal zones.
  There are taken scans with 3Shape Trios4 before surgery, immediately after, then 3 month and 1 year follow up to compare soft tissue stability
The change of position of implant using surgical guide | Before surgery and immediately after surgery
  To compare implant position accuracy using surgical guide, the following two things will be compared: DICOM after the surgery witch contains information on the implant position in the bone and the STL file witch contains information on implant position before the surgery.
  There are taken cone beam computer tomography before and immediately after surgery, then 3 month and 1 year follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Ģirts Šalms, Asoc.prof, Study Director — Riga Stradiņš University
Locations (1):
- Adenta, Riga, Latvija, Latvia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexopoulou M, Lambert F, Knafo B, Popelut A, Vandenberghe B, Finelle G. Immediate implant in the posterior region combined with alveolar ridge preservation and sealing socket abutment: A retrospective 3D radiographic analysis. Clin Implant Dent Relat Res. 2021 Feb;23(1):61-72. doi: 10.1111/cid.12974. Epub 2021 Jan 13. PMID 33438320
- [Background] Sanz-Martin I, Permuy M, Vignoletti F, Nunez J, Munoz F, Sanz M. A novel methodological approach using superimposed Micro-CT and STL images to analyze hard and soft tissue volume in immediate and delayed implants with different cervical designs. Clin Oral Implants Res. 2018 Oct;29(10):986-995. doi: 10.1111/clr.13365. Epub 2018 Sep 23. PMID 30246362
- [Background] Guidetti LG, Monnazzi MS, Piveta AC, Gabrielli MA, Gabrielli MF, Pereira Filho VA. Evaluation of single implants placed in the posterior mandibular area under immediate loading: a prospective study. Int J Oral Maxillofac Surg. 2015 Nov;44(11):1411-5. doi: 10.1016/j.ijom.2015.06.021. Epub 2015 Jul 18. PMID 26194771
- [Derived] Gnusins V, Akhondi S, Zvirblis T, Pala K, Gallucci GO, Puisys A. Chairside vs Prefabricated Sealing Socket Abutments for Posterior Immediate Implants: A Randomized Clinical Trial. Clin Implant Dent Relat Res. 2025 Aug;27(4):e70076. doi: 10.1111/cid.70076. PMID 40692347
- See also: Customized sealing socket abutment (SSA) has been claimed to optimize the peri-implant hard and soft tissues in type 1 implant placement. — https://pubmed.ncbi.nlm.nih.gov/33438320/
- See also: To study the hard and soft tissue volume after placing immediate (IMI) or delayed implants (DLI) with a triangular coronal macro-design (Test/T) or a conventional cylindrical design (Control/C). — https://pubmed.ncbi.nlm.nih.gov/30246362/
- See also: The aim of this study was to evaluate the survival of single dental implants subjected to immediate function. Twelve patients with edentulous areas in the posterior mandible were included in the study. — https://pubmed.ncbi.nlm.nih.gov/26194771/